CLINICAL TRIAL: NCT02560584
Title: A Prospective, Open, Comparative, Within Patient Controlled Multicenter Phase 3 Study of Blue Light Cystoscopy With Cysview and White Light Cystoscopy Using KARL STORZ D-Light C PDD Flexible Videoscope System in Detection of Bladder Cancer in Patients With Bladder Cancer
Brief Title: A Study of Blue Light Flexible Cystoscopy With Cysview in the Detection of Bladder Cancer in the Surveillance Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Photocure (Industry)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PC B308/13
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer
Keywords: Non-muscle invasive bladder cancer; NMIBC; Cysview
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Intervention Model Description: This is a prospective, open, comparative, within-patient controlled Phase 3 multicenter study in patients with bladder cancer. There is a maximum of three study visits for an enrolled patient:
  Visit 1: Screening visit Visit 2: Surveillance cystoscopy in white light (WL) followed by blue light (BL) Visit 3: Operating room (OR) cystoscopy in WL followed by BL for patients with suspicion of recurrence after surveillance cystoscopy.
  Cystoscopy in WL followed by BL is performed in all patients after Cysview instillation. Only patients with suspicious lesions at Visit 2 continue to a second cystoscopy in WL followed by BL at Visit 3.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cysview arm (Experimental): In this single-arm trial, Cystoscopy in white light followed by blue light (BL) is performed in all applicable patients during 2 study visits; Visit 2 (Surveillance) and Visit 3 (Operating room procedure)
  All patients receive instillation of 100 mg hexaminolevulinate hydrochloride as intravesical solution (50 mL) in the bladder prior to cystoscopy. Retention time: 1-3 hours.
  Surveillance cystoscopy is performed with the investigational device KARL STORZ D-Light C PDD Flexible Videoscope System
  Interventions: Drug: Hexaminolevulinate hydrochloride; Device: KARL STORZ D-Light C PDD Flexible Videoscope System

INTERVENTIONS:
Drug: Hexaminolevulinate hydrochloride — Instillation in bladder
  Other Names: Cysview
Device: KARL STORZ D-Light C PDD Flexible Videoscope System — Cystoscopy procedure

SUMMARY:
The purpose of this study is to investigate if blue light cystoscopy with Cysview improves detection of tumors in patients with bladder cancer during surveillance cystoscopy, using the KARL STORZ D-Light C PDD Flexible Videoscope System. Another purpose is to investigate if Cysview and blue light is safe and effective when used repeatedly.

ELIGIBILITY:
1. Patients with bladder cancer in follow-up for tumor recurrence (Note: Patients must be included only at the first surveillance cystoscopy after a histologically confirmed tumor. The histologically confirmed tumor could either be from a TURB or from a surveillance cystoscopy where a biopsy was taken and a tumor was confirmed by histology)
2. History of one or more of the following:

   * Multiple tumors
   * Recurrent tumors
   * High grade tumor(s)

Exclusion Criteria:

1. Gross haematuria. (Note: Gross haematuria is defined as a heavy bladder bleed resulting in significant amounts of blood in the urine, which may visually limit cystoscopy. Where the haematuria is light, the patient should not be excluded, if in the investigator's opinion, rinsing and/or electro-cautery during cystoscopy will alleviate the haematuria limitations to cystoscopy)
2. Patients who cannot undergo in-office or operating room cystoscopy (Note: Training patients are eligible even if they cannot undergo operating room cystoscopy)
3. Patients who have received Bacillus Calmette-Guérin (BCG) immunotherapy or intravesical chemotherapy within the past 6 weeks prior to the procedure
4. Porphyria
5. Known allergy to hexaminolevulinate hydrochloride or a similar compound
6. Pregnancy or breast-feeding (all women of child-bearing potential must document a negative urine pregnancy test before study inclusion and use adequate contraception during the study
7. Participation in other clinical studies with investigational drugs either concurrently or within the last 30 days
8. Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
9. Patients that the investigator believes are unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of participating in the clinical study, uncooperative attitude or unlikelihood of completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schoenberg, MD, Principal Investigator — Montefiore Medical Center; J. Stephen Jones, MD, Principal Investigator — The Cleveland Clinic
Locations (17):
- United States (17):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Langone Urology Associates, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Department of Urology, Chapel Hill, North Carolina
  - Ohio State University The James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma-Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Pohar KS, Patel S, Lotan Y, Trabulsi E, Woods M, Downs T, Huang WC, Jones J, Taylor J, O'Donnell M, Bivalacqua TJ, DeCastro J, Steinberg G, Kamat AM, Resnick MJ, Konety B, Schoenberg M, Jones JS, Daneshmand S; Flexible Blue Light Study Group Collaborators. Safety of repeat blue light cystoscopy with hexaminolevulinate (HAL) in the management of bladder cancer: Results from a phase III, comparative, multi-center study. Urol Oncol. 2022 Aug;40(8):382.e1-382.e6. doi: 10.1016/j.urolonc.2022.04.012. Epub 2022 Jun 22. PMID 35750559
- [Derived] Smith AB, Daneshmand S, Patel S, Pohar K, Trabulsi E, Woods M, Downs T, Huang W, Taylor J, Jones J, O'Donnell M, Bivalacqua T, DeCastro J, Steinberg G, Kamat A, Resnick M, Konety B, Schoenberg M, Jones JS, Lotan Y; Flexible Blue Light Study Group Collaborators. Patient-reported outcomes of blue-light flexible cystoscopy with hexaminolevulinate in the surveillance of bladder cancer: results from a prospective multicentre study. BJU Int. 2019 Jan;123(1):35-41. doi: 10.1111/bju.14481. Epub 2018 Aug 11. PMID 29979488
- [Derived] Daneshmand S, Patel S, Lotan Y, Pohar K, Trabulsi E, Woods M, Downs T, Huang W, Jones J, O'Donnell M, Bivalacqua T, DeCastro J, Steinberg G, Kamat A, Resnick M, Konety B, Schoenberg M, Jones JS; Flexible Blue Light Study Group Collaborators. Efficacy and Safety of Blue Light Flexible Cystoscopy with Hexaminolevulinate in the Surveillance of Bladder Cancer: A Phase III, Comparative, Multicenter Study. J Urol. 2018 May;199(5):1158-1165. doi: 10.1016/j.juro.2017.11.096. Epub 2017 Dec 2. PMID 29203268

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cysview Arm
Started | 304
Completed | 304
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a single-arm trial. All participants received the same intervention. All enrolled participants received Cysview and an examination in the office and were referred to a second procedure in the operating room if medically indicated in the first examination. Baseline characteristics are reported for all enrolled participants.
Arm/Group | Cysview Arm
Number analyzed (Participants) | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 296
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 272
  More than one race | 0
  Unknown or Not Reported | 2
Number of Previous Recurrences [Mean (Standard Deviation); unit: number of previous recurrences] | 1.7 (2.0)
History of CIS [Count of Participants; unit: Participants] | 127
History of High Grade (Grade 2 or 3) Ta or T1 [Count of Participants; unit: Participants] — Under the American Joint Committee on Cancer (AJCC) staging system, also known as the Tumor-Node-Metastases (TNM), pathological stages of NMIBC includes the following: (1) papillary tumors confined to the epithelial mucosa (stage Ta), (2) tumors invading the subepithelial tissue (i.e., lamina propria; T1), and (3) carcinoma in situ. The 1973 World Health Organization (WHO) classification was the widely accepted format for grading bladder neoplasia. The 1973 version designated tumors as either papilloma, grade 1, 2, or 3, whereas the 2004 revision designated tumors as 'low' or 'high' grade.
  Participants | 222
Patients Treated with intravesical chemotherapy [Count of Participants; unit: Participants] | 114
Patients with Previous Treatment with BCG Immunotherapy [Count of Participants; unit: Participants] | 251

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Histologically Confirmed Malignancy Where Malignancy is Only Detected With Blue Light Cystoscopy With Cysview and Not White Light Cystoscopy
Description: In the subsection of patients with histologically confirmed malignancy, the proportion of patients detected only by the use of blue light cystoscopy with Cysview is measured.
Time Frame: At time of cystoscopy procedure
Population: Patients with histologically confirmed malignancy
Measure: Count of Participants; unit: Participants
Arm/Group | Cysview Arm
Number analyzed (Participants) | 63
Participants | 13
Statistical Analysis 1: Comparison: Cysview Arm; The proportion of patients with malignancy detected only with BLC with Cysview was to be analyzed using an exact one-sided test for a single proportion based on the cumulative binomial distribution with a significance level of 2.5%. Null hypothesis: Malignancy is detected with BL only in 0.5% or less of the patients; Test type: Superiority; p < 0.0001, Exact one-sided test for a single propor

2. Secondary Outcome: Proportion of Patients With Adverse Events Considered Causally Related to Cysview and/or Blue Light in the Surveillance Examination Compared With the OR Examination
Time Frame: At time of cystoscopy procedure
Population: This is a within patient control trial, where the white light (WL) cystoscopy was the comparator. Enrolled participants received a WL and blue light (BL) surveillance examination after Cysview instillation. Operating room (OR) cystoscopy in WL and BL was performed for patients with suspicion of recurrence after surveillance cystoscopy.
Measure: Count of Participants; unit: Participants
Groups:
- Surveillance Examination: Patients who received Cysview instillation in the surveillance examination.
- Surveillance + OR Examination: Patients who received a Cysview instillation in both surveillance and OR examinations.
Arm/Group | Surveillance Examination | Surveillance + OR Examination
Number analyzed (Participants) | 304 | 103
Participants | 6 | 3

3. Secondary Outcome: Proportion of Patients With One or More Carcinoma in Situ (CIS) Lesions Detected With Blue Light Cystoscopy With Cysview and None With White Light Cystoscopy
Description: In the subsection of patients with histologically confirmed CIS, the proportion of patients detected only by blue light cystoscopy with Cysview is measured.
Time Frame: At time of cystoscopy procedure
Population: Number of patients with histologically confirmed CIS
Measure: Count of Participants; unit: Participants
Arm/Group | Cysview Arm
Number analyzed (Participants) | 26
Participants | 9
Statistical Analysis 1: Comparison: Cysview Arm; The proportion of patients with one or more CIS lesions detected with BL and none with WL was to be evaluated using an exact binomial test for single proportion with a significance level of 2.5% (one-sided). Null hypothesis: One or more CIS lesions are detected with BLC with Cysview and none with WL in less than or equal to 0.1% of the patients; Test type: Superiority; p < 0.0001, Exact one-sided test for single proporti

ADVERSE EVENTS:
Time Frame: The period of observation in the surveillance examination was defined as the period from instillation of Cysview until the patient left the hospital. The period of observation in the operating room examination was defined as the period from instillation of Cysview until hospital discharge or for a maximum of 24 hours after the instillation if the patient was still at the hospital.
Arm/Group | Cysview Arm
All-Cause Mortality (participants affected / at risk) | 0/304
Serious Adverse Events (participants affected / at risk) | 1/304
Other Adverse Events (participants affected / at risk) | 17/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysview Arm (N=304)
Aspiration, Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cysview Arm (N=304)
Bladder discomfort, Bladder pain, Bladder spasm, Dysuria, Urethral pain, Urinary bladder hemorrhage (Renal and urinary disorders) | 12 (14)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Pain, Pyrexia (General disorders) | 2 (2)
Dermatitis contact, erythema, priuritus (Skin and subcutaneous tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02560584/Prot_SAP_000.pdf